CLINICAL TRIAL: NCT04212585
Title: The Status of Helicobacter Pylori Infection Among Children Visiting Assiut Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebtihal Ramadan Hashem, Principal Investigator, Assiut University
Other Study IDs: H.Pylori status
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with upper gastrointestinal symptoms
  Interventions: Diagnostic Test: Serology test
- children without upper gastrointestinal symptoms
  Interventions: Diagnostic Test: Serology test

INTERVENTIONS:
Diagnostic Test: Serology test — Serology for Helicobacter pylori (immunoglobulin G for all sites, immunoglobulin M optional, immunoglobulin A optional) will be collected from all participants. 90 samples (immunoglobulin G, immunoglobulin M and immunoglobulin A) at least needed from each site.
  Stool antigen for Helicobacter pylori

SUMMARY:
The aim of this study is to estimate the prevalence of Helicobacter pylori infection among Egyptian children attending to healthcare facilitates using different diagnostic tools.

DETAILED DESCRIPTION:
The prevalence of H. pylori infection, which has a ubiquitous distribution, varies depending on socioeco- nomic factors and age. in the context of a decreased trend in H. pylori prevalence, at least 50% of the world's hu-man population are carriers of the microorganism, with a prevalence much higher in developing countries than in developed countries. H. pylori infection was evaluated in 286 Egyptian school children, and the overall prevalence was > 72%. Acquisition of the infection occurs mostly in early childhood; therefore, a better understanding of the epidemiology and the risk factors associated with H. pylori infection in the pediatric population is important to clarify the natural history and complications of the infection and programming eradication strategies.

Currently, little data exist regarding the epidemiology of H. pylori associated infection in our region., especially in children. Therefore, this study aims to determine the prevalence of H. pylori among children.

ELIGIBILITY:
Inclusion Criteria:

* All children (<18 years) attending healthcare facilities for any reason will be enrolled after informed consent of their parents to participate in the study.

Participants will be recruited from the following sources:

1. Children with non-GI symptoms (ophthalmology, ear, nose, and throat , chest departments .. etc)
2. Children with GI symptoms undergoing upper GI endoscopy (from GI endoscopy units).

Simple questionnaire will be used to collect demographic data, socioeconomic status, dietary habits, and gastrointestinal complaints from parents of all participants before testing for Helicobacter pylori.

Exclusion Criteria:

1. Patients refusing to be enrolled in the study.
2. For any diagnostic test other than serology (stool antigen, rapid Urease test, urea breath test, histopathology) the following patients will be excluded:

   * Children received any antibiotics in the last month
   * Children received bismuth compounds in the last month.
   * Children received proton pump inhibitors in the last 2 weeks.
   * Children presenting with upper gastrointestinal bleeding.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Egyptian Children aged from 0 years to 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of H. pylori in children hospital attendees. | 2 years
  We need to estimate prevalence of H.Pylori infection among all children admitted in Assiut University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Magda S Hasan, M.D., Study Director — Assiut University

REFERENCES:
- [Background] Blecker U. Helicobacter pylori-associated gastroduodenal disease in childhood. South Med J. 1997 Jun;90(6):570-6; quiz 577. PMID 9191731
- [Background] Tonkic A, Tonkic M, Lehours P, Megraud F. Epidemiology and diagnosis of Helicobacter pylori infection. Helicobacter. 2012 Sep;17 Suppl 1:1-8. doi: 10.1111/j.1523-5378.2012.00975.x. PMID 22958148
- [Background] Mohammad MA, Hussein L, Coward A, Jackson SJ. Prevalence of Helicobacter pylori infection among Egyptian children: impact of social background and effect on growth. Public Health Nutr. 2008 Mar;11(3):230-6. doi: 10.1017/S1368980007000481. Epub 2007 Aug 1. PMID 17666124
- [Background] Takahashi M, Kimura H, Watanabe K. Helicobacter pylori infection in patients with idiopathic short stature. Pediatr Int. 2002 Jun;44(3):277-80. doi: 10.1046/j.1442-200x.2002.01557.x. PMID 11982896
- [Background] Malaty HM, Logan ND, Graham DY, Ramchatesingh JE, Reddy SG. Helicobacter pylori infection in asymptomatic children: comparison of diagnostic tests. Helicobacter. 2000 Sep;5(3):155-9. doi: 10.1046/j.1523-5378.2000.00024.x. PMID 10971680
- [Background] Roma E, Miele E. Helicobacter pylori Infection in Pediatrics. Helicobacter. 2015 Sep;20 Suppl 1:47-53. doi: 10.1111/hel.12257. PMID 26372825
- [Background] Sustmann A, Okuda M, Koletzko S. Helicobacter pylori in children. Helicobacter. 2016 Sep;21 Suppl 1:49-54. doi: 10.1111/hel.12341. PMID 27531540
- [Background] Plummer M, Franceschi S, Vignat J, Forman D, de Martel C. Global burden of gastric cancer attributable to Helicobacter pylori. Int J Cancer. 2015 Jan 15;136(2):487-90. doi: 10.1002/ijc.28999. Epub 2014 Jun 11. PMID 24889903